CLINICAL TRIAL: NCT01284088
Title: A Prospective, Randomized, Open Label, Trial Comparing the PrePex™ Device to Surgical Circumcision for Rapid Scale Up of Male Circumcision in Resource Limited Settings
Brief Title: Comparing the PrePex™ Device to Surgical Circumcision for Rapid Scale Up of Male Circumcision in Resource Limited Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Rwanda (Other Government)
Responsible Party: Principal Investigator, Agnes Binagwaho M.D., Permanent Secretary of Health, Ministry of Health, Rwanda
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RMC-01
Record Dates: First submitted 2011-01-24; First posted 2011-01-26 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: HIV
Keywords: Male Circumcision; HIV Prevention; Medical Device

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PrePex™ (Experimental): Adult male circumcision by the PrePex™ Device
  Interventions: Device: PrePex™ device for adult male circumcision
- Surgical (Active Comparator): Adult male surgical circumcision
  Interventions: Procedure: Surgical circumcision

INTERVENTIONS:
Device: PrePex™ device for adult male circumcision — The PrePex™ device is designed to enable bloodless male circumcision procedure with no anesthesia and no sutures.
  Other Names: The PrePex Device; PrePex; PrePex™
  Arms: PrePex™
Procedure: Surgical circumcision — The penis will be surgically circumcised according to one of the WHO recommended circumcision methods as described in the Manual for Male Circumcision under Local Anaesthesia Version 2.5C January 2008
  Arms: Surgical

SUMMARY:
The World Health Organization and UNAIDS cite that male circumcision can reduce the lifetime risk of HIV infection by 60% in high risk areas such as Sub Saharan Africa.

Rwanda has a national plan to offer a voluntary circumcision program to 2 million adult men in 2 years as part of a comprehensive HIV prevention package. To achieve this goal, the government is continuing to study the PrePex™ device, developed to enable rapid adult male circumcision in resource limited settings.

The study will enroll one hundred and fifty (150) persons scheduled for voluntary circumcision. The subjects will be randomly divided into two unbalanced study arms, PrePex™ arm which will include about a hundred and twenty (100) subjects and surgical circumcision arm which will include about sixty (50) subjects.

Study duration per subject will be 9 weeks.

DETAILED DESCRIPTION:
The World Health Organization and UNAIDS cite that male circumcision can reduce the lifetime risk of HIV infection by 60% in high risk areas such as Sub Saharan Africa. In 2009, the US Government (USAID) reported that scaling up male circumcision to reach 80 percent of adult and newborn males in 14 African countries by 2015 could potentially avert more than 4 million adult HIV infections between 2009 and 2025 and yield annual cost savings of US$1.4 - 1.8 billion after 2015, with a total net savings of US$20.2 billion between 2009 and 2025.

There are over 38 million adolescent and adult males in Africa that could benefit from male circumcision for HIV prevention. The challenge Africa faces is how to safely scale up a surgical procedure in resources limited settings.

The government of Rwanda has a national plan to decrease the incidence rate of HIV by 50%, and to support this, needs to conduct 2 million voluntary adult male circumcisions in 2 years, a nearly impossible goal with surgical methods. Hence, the government embarked upon a pre-safety and pivotal study to test The PrePex™ System, a new device and methodology for rapid adult male circumcision in resource limited settings. Evidence showed the safety and efficacy of the device, as well as the ability to conduct the procedure with no anesthesia, no blood, no sutures and in a standard consultation room.

The government decided to embark upon a controlled, randomized, two arm study comparing the PrePex™ device with the surgical method to have a broader evidence base to support the findings in the pivotal study.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21 - 54 years
* Subject wants to be circumcised
* Uncircumcised
* Agrees to be circumcised by any of the study methods, PrePex™ or Surgical as will be determined randomly
* Able to understand the study procedures and requirements
* Agrees to abstain sexual intercourse and to keep caution not directly rub the cut area if masturbating, for 8 weeks post removal (9 weeks total).
* Agrees to return to the health care facility for follow-up visits (or as instructed) after his circumcision that may take up to 8 weeks
* Subject able to comprehend and freely give informed consent for participation in this study and is considered by the investigator to have good compliance for the study

Exclusion Criteria:

* Active genital infection, anatomic abnormality or other condition, which in the opinion of the investigator prevents the subject from undergoing a circumcision
* Subject with the following diseases/conditions: phimosis, paraphimosis, warts under the prepuce, torn or tight frenulum, narrow prepuce, hypospadias,epispadias
* Known bleeding/coagulation abnormality, uncontrolled diabetes
* Subject who have an abnormal penile anatomy or any penile diseases
* Subject that to the opinion of the investigator is not a good candidate
* Subject that refuse to have an HIV test
* Subject does not agree to anonymous video and photographs of the procedure and follow up.

Ages: 21 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 217 (Actual)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The study's primary goal is to compare the PrePex™ circumcision procedure with one of the approved WHO methods of surgical circumcision. | 9 weeks
  The primary endpoint is the total operative time of the PrePex™ Device circumcision procedure versus the total operative time of surgical circumcision procedure.

SECONDARY OUTCOMES:
Measured circumcision preparation time. | 9 weeks
  The total preparation time of the PrePex™ Device circumcision procedure versus the total preparation time of surgical circumcision procedure
Pain assessment at key time points | 9 weeks
Clinical adverse event rates | 9 weeks
Patient satisfaction | 9 weeks
Time to complete healing | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Binagwaho, M.D., Principal Investigator — Ministry of Health, Rwanda
Locations (1):
- Nyamata District Hospital, Bugesera District, Nyamata Sector, Rwanda

REFERENCES:
- [Derived] Hohlfeld A, Ebrahim S, Shaik MZ, Kredo T. Circumcision devices versus standard surgical techniques in adolescent and adult male circumcisions. Cochrane Database Syst Rev. 2021 Mar 31;3(3):CD012250. doi: 10.1002/14651858.CD012250.pub2. PMID 33786810
- [Derived] Mutabazi V, Kaplan SA, Rwamasirabo E, Bitega JP, Ngeruka ML, Savio D, Karema C, Binagwaho A. HIV prevention: male circumcision comparison between a nonsurgical device to a surgical technique in resource-limited settings: a prospective, randomized, nonmasked trial. J Acquir Immune Defic Syndr. 2012 Sep 1;61(1):49-55. doi: 10.1097/QAI.0b013e3182631d69. PMID 22739133